CLINICAL TRIAL: NCT05601973
Title: A Multicentre Single-arm Phase II Trial of Amivantamab, Lazertinib Plus Bevacizumab in Patients With EGFR-mutant Advanced NSCLC With Progression on Previous Third-generation EGFR-TKI
Brief Title: Amivantamab, Lazertinib and Bevacizumab in Patients With EGFR-mutant Advanced Non-small Cell Lung Cancer With Progression on Previous Third-generation EGFR-TKI
Acronym: AMAZE-lung
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 18-21; 2021-002337-42 (EudraCT Number)
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: EGFR-mutant advanced non-squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — amivantamab; lazertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Amivantamab (fixed dose of 1750 mg (or 2100 mg, i.v. every 3 weeks, until disease progression, or intolerable toxicity) PLUS Lazertinib (240 mg, orally, once daily, until disease progression or intolerable toxicities) PLUS Bevacizumab (Zirabev® is administered at a dose of 15mg/kg, i.v. every 3 weeks, until disease progression, or intolerable toxicity).
  Interventions: Drug: Amivantamab; Drug: Lazertinib; Drug: Zirabev

INTERVENTIONS:
Drug: Amivantamab — Amivantamab is given at a fixed dose of 1750 mg (if baseline body weight is <80 kg) or 2100 mg (if baseline body weight is ≥80 kg), i.v. every 3 weeks, until disease progression, or intolerable toxicity.
Drug: Lazertinib — Lazertinib is given at a dose of 240 mg, orally, once daily. Treatment with lazertinib continues until disease progression or intolerable toxicities.
Drug: Zirabev — Bevacizumab (Zirabev®) is administered at a dose of 15mg/kg, i.v. every 3 weeks, until disease progression, or intolerable toxicity.

SUMMARY:
AMAZE-lung is a multicenter single-arm phase II trial. The protocol treatment consists of amivantamab, lazertinib and bevacizumab (Zirabev®), given in a three-weekly regimen. The primary objective of the trial is to assess the efficacy of amivantamab and bevacizumab added to continued treatment with the third-generation EGFR-TKI lazertinib, in patients with EGFR-mutant advanced NSCLC, who have been previously treated with a third-generation EGFR-TKI in order to provide data on treatment effect and sample size required for a future phase III trial.

In addition, the safety of the treatment combination will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-squamous NSCLC, stage IIIB/C (not amenable to radical therapy) or stage IV according to 8th TNM classification.
2. Presence of a sensitising EGFR-mutation (only patients with exon 19 deletion and/or L858R are eligible) and documentation of T790M status, tested locally by an accredited laboratory.
3. Radiologically confirmed disease progression on previous treatment with osimertinib or lazertinib.Treatment with osimertinib must have been stopped at least 8 days before enrolment.
4. Achieved objective clinical benefit from osimertinib or lazertinib treatment (e.g., documented PR/ CR or SD for ≥6 months while on osimertinib or lazertinib treatment).
5. Measurable disease as defined according to RECIST v1.1.
6. Age ≥18 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Life expectancy ≥12 weeks.
9. Adequate haematological function:

   * Haemoglobin ≥100 g/L,
   * Absolute neutrophil count (ANC) ≥1.5× 109/L,
   * Platelet count ≥75× 109/L.
10. Adequate renal function:

    - Serum creatinine <1.5× ULN and calculated (Cockcroft-Gault formula) or measured creatinine clearance >45 mL/min.
11. Adequate liver function:

    * ALT and AST ≤3× ULN. If the patient has liver metastases, ALT and AST must be ≤5× ULN.
    * Total bilirubin ≤1.5× ULN. Patients with Gilbert's syndrome are eligible if conjugated bilirubin is within normal limits.
12. Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative pregnancy test (b-human chorionic gonadotropin [b-hCG]) within 5 weeks before enrolment and within 3 days before the first dose of protocol treatment. Women of childbearing potential must use highly effective contraceptive methods.
13. Written IC for trial participation must be signed and dated by the patient and the investigator prior to any trial-related intervention.

Exclusion Criteria:

1. Patients with known small cell lung carcinoma (SCLC) transformation.
2. Patients with symptomatic brain metastases. Patients with asymptomatic or previously treated and stable brain metastases may participate in this study. Patients who have received definitive radiotherapy or surgery for symptomatic or unstable brain metastases and have been clinically stable and asymptomatic for at ≥2 weeks before enrolment are eligible, provided they have been either off corticosteroid treatment or are receiving low-dose corticosteroid treatment (≤10 mg/day prednisone or equivalent) for at least 2 weeks prior to enrolment.
3. Patients with an active or past medical history of leptomeningeal disease.
4. Patients with untreated spinal cord compression. Patients who have been definitively treated with surgery or radiotherapy and have a stable neurological status for ≥2 weeks prior to enrolment are eligible provided they are off corticosteroid treatment or are receiving low-dose corticosteroid treatment ≤10 mg/day prednisone or equivalent.
5. Patients with unresolved adverse events (other than alopecia) from prior anticancer therapy that have not resolved to grade ≤1 or baseline.
6. Patients with positive hepatitis B (hepatitis B virus [HBV]) surface antigen (HBsAg) test.
7. Patients with positive hepatitis C antibody (anti-HCV) test.
8. Patients with other clinically active infectious liver disease.
9. Patients who are known positive for HIV, with one or more of the following:

   * Receiving antiretroviral therapy (ART) that may interfere with study treatment
   * CD4 count <350 at screening.
   * AIDS-defining opportunistic infection within 6 months before enrolment.
   * Not agreeing to start ART and be on ART >4 weeks plus having HIV viral load <400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV is under control).
10. Patients with active cardiovascular disease including, but not limited to:

    * Medical history of deep vein thrombosis or pulmonary embolism within 1 month prior to enrolment or any of the following within 6 months prior to enrolment: Myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome.
    * Prolonged corrected QTcF >470 msec, clinically-significant cardiac arrhythmia (e.g., atrial fibrillation with uncontrolled rate) or abnormalities in conduction or morphologiy of electrocardiogram (ECG) (e.g., complete left bundle branch block, third- or second-degree heart block, PR interval >250 msec), or electrophysiologic disease (eg, placement of implantable cardioverter defibrillator).
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years in first degree relatives or any concomitant medications known to prolong QT interval or induce TdP.
    * Uncontrolled (persistent) hypertension: systolic blood pressure >160 mm Hg; diastolic blood pressure >100 mm Hg.
    * Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalisation for CHF (any NYHA class) within 6 months before enrolment.
    * An active or past medical history of pericarditis, pericardial effusion that is clinically unstable, or myocarditis.
    * Pericardial effusion considered due to the disease under study is permitted if clinically stable at screening.
    * Baseline LVEF either <50% or below the lower limit of normal (LLN) per institutional guidelines, as assessed by screening echocardiogram (ECHO) or multigated acquisition (MUGA) scan.
11. Patients with interstitial lung disease (ILD), including drug-induced ILD or radiation pneumonitis.
12. Patients with a history of haemoptysis (≥2.5 mL of bright red blood per episode) within 1 month prior to enrolment.
13. Patients with evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation).
14. Patients with current or recent (within 10 days before enrolment) use of aspirin (>325 mg/day) or treatment with dipyridamole, ticlopidine, clopidogrel, and clostazol.
15. Patients with current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for >2 weeks prior to enrolment.

    * The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to enrolment.
    * Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR <1.5× ULN and aPTT is within normal limits within 14 days prior to enrolment.
    * Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
16. Patients with serious, non-healing wound, active ulcer, or untreated bone fracture.
17. Patients who had a core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to enrolment.
18. Patients who had major surgery or significant traumatic injury within 28 days prior to enrolment.
19. Patients who had placement of a vascular access device within 2 days prior to prior to enrolment.
20. Patients with a history of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to enrolment.
21. Patients with clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding.
22. Patients with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
23. Patients with concurrent or prior malignancy other than the disease under study.

    Some exceptions require consultation with the ETOP IBCSG Partners
24. Patients with uncontrolled illness, including but not limited to:

    * Uncontrolled diabetes.
    * Ongoing or active infection, or diagnosed or suspected viral infection.
    * Active bleeding diathesis.
    * Impaired oxygenation requiring continuous oxygen supplementation.
    * Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated drug, or previous significant bowel resection
    * Psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements.
    * Any ophthalmologic condition that is clinically unstable.
25. History of hypersensitivity to either the drug substance or any excipients in amivantamab, lazertinib and/ or bevacizumab.
26. Prior chemotherapy for NSCLC.
27. Prior treatment with bevacizumab or another anti-angiogenic inhibitor.
28. Prior treatment with a MET/EGFR-targeting antibody.
29. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
30. Women who are pregnant or in the period of lactation.
31. Women of childbearing potential or men who are sexually active with a woman of childbearing potential, who are not willing to use at least one method of highly effective contraception while receiving protocol treatment and for at least 6 months after the last dose of protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of amivantamab and bevacizumab added to continued treatment with a third-generation EGFR-TKI (osimertinib or lazertinib) | from date of enrolment until 12 weeks of follow-up.
  The primary endpoint to assess the efficacy of amivantamab and bevacizumab added to continued treatment with a third-generation EGFR-TKI (osimertinib or lazertinib) is the objective response rate (ORR), investigator assessed, at 12 weeks according to RECIST v1.1. ORR is defined as the rate of patients, among all enrolled patients, that achieve a best overall response [complete response (CR) or partial response (PR)] across all post-enrolment tumour-assessment time-points.

SECONDARY OUTCOMES:
To evaluate secondary measures of clinical efficacy including progression-free survival (PFS), overall survival (OS), duration of response (DoR), disease control rate (DCR). | from date of first documented objective response (CR or PR) to the date of first documented progression/relapse or death, assessed up to 24 months.
  Secondary endpoint: Duration of response (DoR)
To evaluate secondary measures of clinical efficacy including progression-free survival | time from enrolment date until documented progression or death or date of last tumour assessment (for patient without PFS), assessed up to 24 months
  Secondary endpoint: Progression-free survival (PFS) according to RECIST v1.1
To evaluate secondary measures of clinical efficacy including progression-free survival | from date of enrolment until 12 weeks after enrolment.
  Secondary endpoint: Disease control rate (DCR) according to RECIST v1.1 patients, among all enrolled patients, that achieve CR or PR or disease stabilisation at 12 weeks.
To evaluate secondary measures of clinical efficacy including progression-free survival | from date of enrolment until death from any cause. Censoring will occur at the last follow-up date (appr. 24 months after FPI).
  Secondary endpoint: Overall survival (OS)
Safety and tolerability of the treatment based on any reported adverse events (any-cause, treatment-related, AEs leading to dose interruptions, withdrawal of treatment, and death as well as severe, serious and selected adverse events) and deaths | From first patient enrolled until last patient last visit (about 24 months after FPI).
  Secondary endpoint: Safety and tolerability (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Soo, MD FRACP, Study Chair — National University Hospital, Singapore
Locations (18):
- France (3):
  - Chu Angers, Angers
  - Centre Hospitalier d'Avignon, Avignon
  - Centre Léon Bérard, Lyon
- AO SM Misericorida Perugia, Perugia, Italy
- Netherlands Cancer Institute (NKI), Amsterdam, Netherlands
- Spain (8):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario Alicante Dr Balmis ISABIAL, Alicante
  - ICO Badalona, Badalona
  - Vall d´Hebron University Hospital VHIO, Barcelona
  - Hospital Universitario Basurto, Bilbao
  - Catalan Institute of Oncology, L'Hospitalet de Llobregat
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital clínico universitario de Valladolid, Valladolid
- Switzerland (4):
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Universitätsklinik für Medizinische Onkologie, Inselspital, Bern
  - Hôpitaux universitaires de Genève (HUG), Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP